CLINICAL TRIAL: NCT00127725
Title: A Double Blind Randomised Controlled Trial of Pulsed Electromagnetic Field (PEMF) Stimulation in Acute Tibial Shaft Fractures
Brief Title: Pulsed Electromagnetic Field (PEMF) Stimulation for Tibia Fractures
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sydney South West Area Health Service (Other Government)
Collaborators: Biomet Australia Pty Ltd. (Industry); St George Hospital, Australia (Other); South West Sydney Local Health District (Other); University of Wollongong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/023
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-08

CONDITIONS: Tibial Fractures
Keywords: tibia; fracture; PEMF; electromagnetic; non-union; revision; Diaphyseal fractures of the tibia
MeSH Terms: conditions — Tibial Fractures; Fractures, Bone

INTERVENTIONS:
Device: Pulsed electromagnetic field stimulation

SUMMARY:
Fractures of the tibial shaft (diaphysis) are some of the most common long bone fractures. They most frequently occur in males less than 40 years of age. Despite advancements in the surgical management of these fractures, the precarious blood supply and lack of soft-tissue cover of the shaft of the tibia make these fractures vulnerable to non-union and infection. These complications often require multiple procedures, extended time off of work, and can result in ongoing poor mobility. This is reflected in the surgical revision rate that the scientific literature has recorded as being between 20 and 30%.

Pulsed electromagnetic field (PEMF) stimulation has been shown to be a safe and effective treatment for non-unions of the tibia. These are fractures in which the bone has failed to unite and the healing process has ceased. The PEMF is delivered via a device such as the EBI Bone Healing System®, which straps onto the limb overlying the fracture. It is lightweight and portable using a rechargeable battery for power. It is compatible with internal and external fixation and may also be worn over a plaster or fibreglass cast. It is usually kept in place for ten hours per day and used for a period of three months or until the fracture unites. In animal models, PEMF stimulation has been demonstrated to improve the time to fracture healing in acute fractures. There have been no demonstrated side effects of the therapy.

The study hypothesis is that PEMF stimulation during the first twelve weeks after fracture, in addition to normal surgical care, will increase the union rate for these fractures and thereby significantly reduce the surgical revision rate within the first twelve months following fracture.

DETAILED DESCRIPTION:
Study Objectives:

This is a randomized controlled study whose objective is to determine whether PEMF stimulation as an adjunct therapy has a clinically significant effect on the morbidity associated with tibial shaft fractures.

It is a two-armed study. The active treatment arm involves participants with acute tibial shaft fractures who have been randomized to receive a PEMF stimulation device to be worn over the fracture site for 10 hours per day during the first twelve weeks after injury. The control arm involves participants with acute tibial shaft fractures who have been randomized to receive a placebo device to be worn over the fracture site for 10 hours per day during the first twelve weeks after injury.

Primary Aim:

* To determine whether the use of a PEMF stimulation device as adjunct therapy for acute tibial shaft fractures reduces the surgical revision rate in the 12 months after injury.

Revision surgery for the purposes of this study is defined as any surgery on the injured leg (between the knee joint and ankle joint) more than 14 days after the accident, except operations designed to provide initial skin coverage or skin closure, or the removal of an external fixateur as an isolated procedure. Revision surgery will be classified as minor or major. Minor revision will be defined as dynamisation of an intramedullary nail through the percutaneous removal of a static locking screw. Major revision surgery will include all other revision surgery as defined above. Major revision surgery will be sub-classified as procedures involving either bone grafting, and/or revision of fixation, and/or for the treatment of established infection, or amputation, and the rates will be compared across treatment and placebo arms.

Secondary Aims:

* To determine whether the use of a PEMF stimulation device as adjunct therapy for acute tibial shaft fractures increases the radiological and clinical union rates at 12, 26 and 52 weeks after injury. A fracture will be deemed to have radiologically united at these times if by independent observation, two orthopaedic consultants agree that three bony cortices are bridged by bony callus on an anteroposterior and lateral plain X-ray at these times. If the two reviewers disagree, a third opinion will be sought which will be final. A fracture will be deemed to have clinically united if it is deemed stable under clinical examination by the treating orthopaedic surgeon at these times.
* To determine whether the use of a PEMF stimulation device as adjunct therapy for acute tibial shaft fractures increases the patients' general health score, as measured by the SF-36 general health survey; and function of the injured limb, as measured by the Lower Extremity Functional Scale at 12, 26 and 52 weeks after injury.

Primary Hypothesis:

* That there will be significantly lower rates of surgical revision within 12 months of injury in those participants who received active PEMF stimulation for the first 12 weeks after injury.

Secondary Hypotheses:

* That there will be increased union rates at 12, 26 and 52 weeks after fracture among participants who received active stimulation.
* That the average score on a general health survey and region specific health survey will be higher among participants who received active stimulation.

Research Plan

Study Population:

All adults (18 years and over) with diaphyseal fractures of the tibia who present to a recruiting hospital during the study period will be eligible to enrol into the study. The AO classification 42 will be used to define tibial shaft fractures. Any fracture that extends into the articular surface will be excluded. From an analysis of previous Liverpool patients and the literature, the investigators expect that this population will be 75% - 85% male with an average age of 30-35 years old. There will be no upper limit to ages. If a participant has sustained bilateral tibial shaft fractures, each will be enrolled separately, left before right.

Eligible patients will be approached by a senior member of their treating team, either registrar or consultant, and given an information sheet to read and have the opportunity to have any questions answered. They will then be asked to sign a consent form if they would like to participate in the study. Interpreters will be used during this process for non-english speaking patients.

There will be a 14-day window period post injury in which the device must be applied for the patient to enter the study. If there is any reason why the device cannot be applied by this time, the patient will be excluded from the study. The most commonly encountered reason the investigators expect for this will be a patient who remains in an Intensive Care Unit over 14 days, where electrically sensitive equipment is being used for patient care.

Patients with pacemakers or defibrillators will be excluded, as PEMF stimulation may affect some types of these devices. Patients with pathological fractures due to malignant tumours will be excluded. Pregnant patients will be excluded, as the device is yet to be studied in pregnancy. Patients without the cognitive ability to consent are excluded.

The recruiting hospitals are Liverpool Hospital, St. George Hospital, Westmead Hospital, Nepean Hospital and Wollongong Hospital. Approval has been granted for the study to commence through each hospital's Human Research Ethics Committee. Recruitment of patients will commence on Monday August 14, 2005, at each of these hospitals. Recruitment will end after the target of 340 participants has been enrolled into the study.

Baseline Measures:

Participants will be asked to complete a brief questionnaire on enrolment to determine potential risk factors for non-union. These data will be that of age, smoking, general medical conditions and medications used. The participants' current occupation will also be sought as this may effect the time taken for return to work.

The treating doctor will be asked to complete a questionnaire on other risk factors. This will include details of the mechanism of injury, whether the injury was open or closed (and the Gustillo grade of an open injury), other injuries the participant has sustained, and the treatment received for their injuries, as well as the patients' insurance status. The definitive treatment for the tibia fracture will be classified as either external fixation with casts (plater of paris or fibreglass), intramedullary nailing, internal fixation with plates and screws, or external fixation.

Copies of the initial X-rays will be collected. The fractures will be classified into the nine fracture patterns as defined under the AO classification system by a panel of three orthopaedic consultants experienced in trauma.

Randomisation Process:

After the consent form has been signed and the baseline data collected, the participants will be assigned to either active or inactive arms by the NH&MRC Clinical Trials Centre (CTC) located at Sydney University. Devices will come from a pool of seventy devices, which have been supplied by BiometÒ Australia and are commercially known as the EBI Bone Healing System®. Thirty-five of these devices will be active and thirty-five inactive, and they will be randomly numbered from 1 to 70 by the CTC. The CTC will have the code for active and inactive devices and will conduct the randomisation process using the statistical technique of minimisation, a dynamic allocation process designed to balance known risk factors across treatment arms. The two factors that will be minimised for are the recruiting hospital and whether the injury was closed or open. A device will then be randomly assigned from the available pool of either active or inactive devices, and this assigned device will then be fitted to the patient. The researchers, company representatives, surgeons and patients will all remain blinded to active/inactive arms until all the data have been collected and analysed.

Interventions:

Enrolment in the study will not affect any other aspect of the participants' care. All participants will undergo the normal surgical intervention and follow up for their tibial shaft fracture and any other injuries as recommended by their treating surgeons.

After a participant has been assigned with a device number, sales representatives of BiometÒ Australia will fit them with it within three working days, in either the hospital ward or the participant's home. Participants will receive instructions on how to use the device, and be required to wear the device for ten hours per day for a period of twelve weeks. The devices are manufactured to record the amount of time in which they have been used and thereby measure compliance. Non-compliance will be defined as average use of less than six hours per day. Participants will also be asked at twelve weeks about their average use of the device.

After twelve weeks the research team or company representatives will collect the devices, replace the straps, clean and check them before they re-enter the pool of devices for assignment.

Data Collection:

Data will be collected at 12, 26, and 52 weeks from both participants and their treating surgeons. Participants will receive a survey in the mail, and then be contacted over the phone to attain their answers. On each occasion they will be asked whether they have had any further procedures on their leg, and if so at which hospital and by whom. At three months they will also be asked about their average use of the device, whether they are seeing their surgeon in private rooms or a hospital clinic and of their insurance status. That is, are they being treated under medicare, private health insurance, workers compensation, or third party insurance. They will be asked if they have managed to return to work, and to complete the Lower Extremity Functional Score as well as the Short Form-36 (a general health survey). The phone questionnaire is expected to take 15-30 minutes each time.

Their surgeons will also be contacted at 12, 26 and 52 weeks to determine if there has been any further surgery or other complications, and to gain their opinion on fracture union. Copies of their routine pre-operative and twelve week X-rays will be collected for review. Preoperative X-rays will be classified according to the AO classification system into the 9 sub classifications of tibial shaft fractures by a panel of three orthopaedic surgeons. Two orthopaedic surgeons experienced in trauma, who will remain blinded to the treatment arm of the patients, will assess the twelve-week X-rays to determine if union has occurred. Fracture union rates at twelve weeks will be quantified. Fracture union will be defined as mature callus bridging in three of four cortices over the fracture site on two radiographic views. If there is disagreement amongst the two surgeons, the X-rays shall be reviewed by a third surgeon whose opinion shall be final. For fractures that have failed to unite at twelve weeks, their surgeons will be contacted to determine union rate at six months and their plain X-rays will be collected and reviewed. If they have undergone any surgery, their medical records and operation reports will be examined to determine the reason for the surgery and the exact operation undergone. This is to ascertain surgical revision rate and union rate at 12, 26 and 52 weeks post injury.

Potential Significance:

If shown to be effective, this device may become a common adjunct to the management of tibia fractures and significantly decrease the rate of revision surgery and increase the rate of union seen with these fractures. It may also be considered for use in other long bone fractures.

ELIGIBILITY:
Inclusion Criteria:

* Acute diaphyseal fracture of the tibia (AO classification 42)

Exclusion Criteria:

* Pathological fracture secondary to tumours.
* Pregnant patients.
* Patients with permanent pacemakers or defibrillators.
* If the device is unable to be applied by 14 days post fracture.
* Patients who lack the cognitive ability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340
Dates: Start 2005-08; Study Completion 2009-08

PRIMARY OUTCOMES:
Surgical revision rate in the 12 months after fracture

SECONDARY OUTCOMES:
Fracture union rate at 12, 26 and 52 weeks after fracture
General health score and lower extremity functional score at 12, 26 and 52 weeks after fracture

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Harris, MBBS, Principal Investigator — Sydney South West Area Health Service; Hamish C Rae, MBBS, Principal Investigator — Sydney South West Area Health Service
Locations (5):
- Australia (5):
  - Westmead Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Nepean hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales